CLINICAL TRIAL: NCT02134249
Title: Diosmin Versus Cabergoline for Prevention of Ovarian Hyperstimulation Syndrome
Acronym: infertility
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid abd aziz mohamed, lecturer of ob/gyn, Benha University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: khalid-ahmed
Record Dates: First submitted 2014-05-04; First posted 2014-05-09 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Infertility
Keywords: infertility; ICSI; OHSS; Diosmin; Cabergoline
MeSH Terms: conditions — Infertility | interventions — Diosmin; Cabergoline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Diosmin group) (Active Comparator): In group A, (Diosmin group), 2 tab / 8 hs Diosmin ( 500mg) will be given from at day of HCG injection and for 14 days.
  Interventions: Drug: Diosmin
- Group B(Cabergoline group) (Active Comparator): while in group B (Cabergoline group), 1 tab/day Cabergoline(Dostinex)( 0.5 mg) will be given at day of HCG injection and for 8 days .
  Interventions: Drug: Cabergoline

INTERVENTIONS:
Drug: Diosmin — 2 tab / 8 hs Diosmin ( 500mg) will be given at day of HCG injection and for14 days
  Other Names: Daflon
  Arms: Group A (Diosmin group)
Drug: Cabergoline — 1 tab/day Cabergoline( 0.5 mg) will be given at day of HCG injection and for 8 days
  Other Names: Dostinex
  Arms: Group B(Cabergoline group)

SUMMARY:
The purpose of this study is to compare the effect of oral Diosmin to oral Cabergoline in the prevention of ovarian hyperstimulation syndrome (OHSS) in high-risk women underwent intracytoplasmic sperm injection (ICSI).

DETAILED DESCRIPTION:
Two hundred women at risk of ovarian hyperstimulation syndrome during ICSI cycles will be randomly scheduled into two equal groups. In group A, (Diosmin group), 2 tab / 8 hs Diosmin ( 500mg) will be given at day of HCG injection and for 2 weeks ; while in group B (Cabergoline group), 1 tab/day Cabergoline( 0.5 mg) will be given at day of HCG injection and for eight days.

ELIGIBILITY:
Inclusion Criteria: infertile women undergoing intracytoplasmic sperm injection or polycystic ovarin syndrome (PCO) with one of the following:

1. Presence of more than 20 follicles by ultrasound
2. E2 more than 3000 pg/ml
3. Retrieval of more than 15 follicles

Exclusion Criteria:

* none

Ages: 23 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with ovarian hyperstimulation syndrome (OHSS) | every week for eight weeks
  Diagnosis of OHSS was made according to the criteria of Golan et al.. Mild OHSS was classified as: Grade 1 (abdominal distension and discomfort) and Grade 2 (features of grade 1 plus nausea, vomiting and/or diarrhea; ovaries are enlarged from 5 to 12 cm), moderate OHSS as Grade 3 (features of mild OHSS plus ultrasonic evidence of ascites), severe OHSS as Grade 4 (features of moderate OHSS plus evidence of ascites and/or hydrothorax and breathing difficulties) and Grade 5 (all of the above, plus change in the blood volume, increased blood viscosity due to hemoconcentration, coagulation abnormality, and diminished renal perfusion and function).

SECONDARY OUTCOMES:
pregnancy rate | 14 days after embryos transfer
  β-hCG (serum hCG test) will be checked 14 days after embryos transfer

CONTACTS AND LOCATIONS:
Overall Officials: khalid mohamed, MD, Principal Investigator — Department of Obstetrics and Gynecology, Benha University Hospital; ahmed samy, MD, Principal Investigator — Department of Obstetrics and Gynecology, Benha University Hospital
Locations (2):
- Egypt (2):
  - Banha Universty, Banhā, El Qalubia
  - Benha univesity hospital, Banhā, El Qualyobia

IPD SHARING:
Plan to Share IPD: Yes
with other researcher on research gate

REFERENCES:
- [Derived] Tang H, Mourad SM, Wang A, Zhai SD, Hart RJ. Dopamine agonists for preventing ovarian hyperstimulation syndrome. Cochrane Database Syst Rev. 2021 Apr 14;4(4):CD008605. doi: 10.1002/14651858.CD008605.pub4. PMID 33851429